CLINICAL TRIAL: NCT02934139
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of N91115 in Healthy Subjects
Brief Title: MAD Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Cavosonstat (N91115) in Healthy Subjects (SNO-9)
Acronym: (SNO-9)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N91115-1HS-08
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cystic Fibrosis
Keywords: N91115; Cavosonstat; Healthy Volunteer
MeSH Terms: conditions — Cystic Fibrosis | interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cavosonstat (N91115) 400 mg (Experimental): Every 12 hour oral dosing of N91115 for 7 days
  Interventions: Drug: Cavosonstat
- Cavosonstat (N91115) 600 mg (Experimental): Every 12 hour oral dosing of N91115 for 7 days
  Interventions: Drug: Cavosonstat
- Cavosonstat (N91115) 1200 mg (Experimental): Once daily oral dosing of N91115 for 7 days
  Interventions: Drug: Cavosonstat
- Cavosonstat (N91115) 800 mg (Experimental): Every 12 hour oral dosing of N91115 for 7 days
  Interventions: Drug: Cavosonstat
- Placebo (Placebo Comparator): Matched placebo. Oral dosing every 12 hour or once daily for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cavosonstat — CFTR modulator that stabilizes CFTR
  Other Names: N91115
  Arms: Cavosonstat (N91115) 1200 mg; Cavosonstat (N91115) 400 mg; Cavosonstat (N91115) 600 mg; Cavosonstat (N91115) 800 mg
Other: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The present study is designed to assess the safety and tolerability of escalating, multiple ascending doses of Cavosonstat (N91115) in healthy subjects.

DETAILED DESCRIPTION:
This study will assess the safety and tolerability of escalating, multiple ascending doses of Cavosonstat (N91115) in healthy subjects.

Approximately 5 ascending cohorts are planned with approximately 8 subjects per cohort (6 active, 2 placebo). Each subject will undergo screening (Day -28 to Day -2) and, if eligible, return to the unit on Day -1 when eligibility will be reconfirmed.

Eligible subjects will be randomized in a 3:1 ratio to receive investigational medicinal product (IMP) N91115 (daily [QD] or every 12 hours [Q12H]) or matching placebo (QD or Q12H) for 7 days and will be followed for safety while housed in the clinical research unit (CRU) until discharge on Day 8. Pharmacokinetics will be followed from Study Day 1 through the morning of Study Day 8. The subjects will be discharged from the CRU and complete the post treatment withdrawal phase, including a follow-up phone call on Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Healthy, determined at the screening medical evaluation (including but not limited to medical history, physical examination, and clinical laboratory evaluations)
3. Male or female, between 18 and 55 years of age, inclusive at screening
4. Caucasian (as reported by patient)
5. The following applies to female subjects:

   1. Negative serum pregnancy test (for women of child-bearing potential) at screening and negative urine pregnancy at Day -1
   2. Willing to use at least 1 highly effective method of birth control (excluding hormonal contraceptives) after signing consent, including abstinence which must be in use from the time of consent through the 30 days after completing the double-blind study drug
6. The following applies to male subjects:

   1. Agrees to use a condom or abstinence, and agrees to refrain from sperm donation from date of informed consent signing through the 30 days after completing the double-blind study drug or
   2. Has documentation of azoospermia or vasectomy
7. Non-smoker (or other nicotine user) as determined by history (no nicotine use over the past 6 months) and a negative cotinine test at screening and Day -1
8. Body mass index between 18 and 32 kg/m2 inclusive at screening, and weighs at least 50 kg at screening
9. No clinically significant vital sign findings including no clinically significant abnormal findings related to their systolic or diastolic BP at screening or prior to dosing on Day 1, per the investigator's judgment.
10. No clinically significant abnormal findings in 12-lead ECG, per the investigator's judgment, at screening or prior to dosing on Day 1
11. No clinically significant abnormalities in hematology, clinical chemistry, and urinalysis results that would interfere with the study assessments at screening

Exclusion Criteria:

1. History of any illness or condition that in the opinion of the investigator could confound the results of the study or pose additional risk when administered IMP, such as clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the investigator or designee
2. Concurrent disease or condition, that, in the opinion of the investigator, would make the subject unsuitable for participation in the clinical study
3. Any of the following findings on a 12-lead ECG done at screening:

   1. HR < 45 bpm or > 95 bpm
   2. QTcF > 450 msec for males and >470 msec for females
   3. PR > 220 msec
   4. QRS duration > 110 msec
   5. ST segment abnormal
   6. T-wave changes
   7. QRS, ST, or T-wave findings making it technically difficult to determine the QT intervals
4. Any of the following on 24-hour ambulatory ECG (Holter) monitoring at screening:

   a. Supraventricular ectopy i. Singlets: > 200 / 24 hours ii. Couplets: > 20 / hour iii. Runs: > 10 beats b. Ventricular ectopy i. Unifocal singlets: > 100 / 24 hours ii. Unifocal couplets: > 20 / hour iii. Complex of multifocal singlets: > 50 / 24 hours iv. Complex of multifocal couplets: > 10 / 24 hours v. Any Run (ventricular tachycardia) c. Heart rate i. < 40 bpm for 1 minute while awake ii. < 35 bpm for 3 minutes while asleep iii. > 120 bpm for 3 minutes (when not exercising) iv. Pauses > 2000 msec d. 2nd or 3rd degree AV block e. Intraventricular conduction delay (IVCD) with QRS duration > 120 msec or right bundle branch block (RBBB) or left buddle branch block (LBBB) other than rare RBBB f. Atrial flutter or atrial fibrillation regardless of rate
5. Disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs as determined by the investigator
6. History of alcohol abuse or drug abuse (including cannabis, cocaine, and opioids) in the year prior to screening
7. Positive alcohol test at screening or Day -1.
8. Positive drug test (including but not limited to cocaine, amphetamines, barbiturates, opiates, benzodiazepines) at screening or Day -1.

   a. A positive drug test for cannabinoids at screening will be allowed if the subject agrees to abstain from use of all forms of cannabinoids during screening and throughout the study and has a negative test at Day -1
9. Positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.
10. Unwilling to limit consumption of coffee and caffeine-containing foods and beverages from Day -1 until discharge on Day 8.
11. Unwilling to avoid use of alcohol or alcohol-containing foods, medications, or beverages from Day -1 until discharge on Day 8.
12. Subject has donated blood (> 500 mL) or blood products within 56 days prior to Day -1.
13. Use of vitamins from Day -7 until end-of-study follow up call, and use of over-thecounter (OTC) medications, prescription medications, or herbal remedies from Day - 14 until end-of-study follow-up call. By exception, acetaminophen ≤ 1000 mg/day is permitted except within 48 hours prior to Day -1. Hormone replacement therapy (HRT) and hormonal contraception is allowed throughout the study. The Medical Monitor and Principal Investigator may allow certain OTC medications by exception if they are not likely to affect study conduct and output.
14. Use of an investigational drug within 30 days prior to Day 1 dosing.
15. Unwilling to abstain from vigorous exercise from Day -1 until discharge on Day 8.
16. Problems understanding the protocol requirements, instructions and study related restrictions, the nature, scope, and possible consequences of the clinical study.
17. Unlikely to comply with the protocol requirements, instructions, and study related restrictions; e.g., uncooperative attitude, unavailable for follow-up call, and/or improbability of completing the clinical study.
18. History of bleeding disorders (i.e., severe hemorrhage, melena, rectal bleeding, nosebleeds, bruising, etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 14 days
  Safety assessments based on clinical evaluations, laboratory assessments, and adverse events

SECONDARY OUTCOMES:
Pharmacokinetic parameters of N91115 and metabolites (Amount of analyte excreted in the urine [Ae]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in urine.
Pharmacokinetic parameters of N91115 and metabolites (% analyte excreted in the urine [Fe]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in urine.
Pharmacokinetic parameters of N91115 and metabolites (area under the curve [AUC]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (maximum concentration [Cmax]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (clearance [CL]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in urine and plasma.
Pharmacokinetic parameters of N91115 and metabolites (accumulation index [Racc]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (Terminal elimination half-life [t1/2]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (time of maximum concentration [Tmax]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (metabolite to parent exposure ratio [M/P ratio]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.
Pharmacokinetic parameters of N91115 and metabolites (terminal elimination rate constant [lambda z]) | 7 days
  Pharmacokinetic parameter of N91115 and metabolites will be measured in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Williams, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No